CLINICAL TRIAL: NCT01825369
Title: Phase 1 Study of the Safety and Pharmacokinetics of Perioperative IV L-carnitine Administration in Patients With Congenital Heart Disease With Increased Pulmonary Blood Flow
Brief Title: Aberrations in Carnitine Homeostasis in Congenital Heart Disease With Increased Pulmonary Blood Flow
Acronym: L-carn
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Changes to cardiac surgery program
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FinemanCarnitine
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Heart Septal Defects, Ventricular; Atrioventricular Septal Defect
Keywords: congenital heart disease; ventricular septal defect; atrioventricular septal defect; increased pulmonary blood flow; nitric oxide
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Atrioventricular Septal Defect; Heart Defects, Congenital | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV L-carnitine (Experimental): L-carnitine (25, 50, or 100mg/kg IV) will be given, 30-60 minutes prior to the initiation of CPB, and a second dose ~2 hr. following separation from CPB (with a minimum of 4 hrs from initial dose). The first 5 subjects will receive 25 mg/kg, with an escalation of dose after each 5 subjects enrolled. The study drug will be brought to the operating room and administered over 5 minutes by the anesthesiologist after an IV has been placed. Prior to the administration of the study drug, and again 24 and 48 hrs after CPB, 3.0 ml of blood will be collected for determinations of carnitine levels (free, total, and acylcarnitine), mitochondrial function, ROS and bioavailable NO as described in Aim 3A. Additional blood (0.5-1.0 ml) will be obtained to determine carnitine levels before CPB, and then before and 0.5, 1.5, 3, 5, 9, 12, and 24h after the second dose.
  Interventions: Drug: IV L-carnitine

INTERVENTIONS:
Drug: IV L-carnitine — See arm description

SUMMARY:
Infants with congenital heart disease and increased pulmonary blood flow have altered carnitine homeostasis that is associated with clinical outcomes; and L-carnitine treatment will attenuate these alterations and improve clinical outcomes.

The investigators will pilot a trial assessing the safety and pharmacokinetics of perioperative IV L-carnitine administration in these patients. To this end, a pilot clinical trial is proposed. Infants with ventricular septal defects or atrioventricular septal defects undergoing complete surgical repair will receive L-carnitine (25, 50, or 100 mg/kg, IV) just prior to cardiopulmonary bypass (CPB) and 2hr after CPB. Carnitine levels will be measured before CPB, and before and 0.5, 1.5, 3, 5, 9, 12, and 24h after the second dose. The safety, pharmacokinetic profile, feasibility, and effect of L-carnitine administration on biochemical parameters, as well as clinical outcomes will be determined. The investigators expect this pilot to provide the data needed to proceed with a placebo-based randomized, controlled, trial.

DETAILED DESCRIPTION:
AIM: To pilot a trial assessing the safety and pharmacokinetics (PK) of perioperative IV L-carnitine administration in these patients. To this end, a pilot clinical trial is proposed. Infants with VSD or AVSD undergoing complete repair will receive L-carnitine, in one of 3 doses (25, 50, or 100 mg/kg, IV), just prior to CPB, and again 2 hr after CPB. Serial blood samples will be obtained to determine free, total, and acylcarnitine levels, and plasma markers of mitochondrial function, oxidative stress, and bioavailable NO. Adverse events will be sought, and clinical outcomes will be assessed.

Study design: The inclusion and exclusion criteria are as described in Aim 3A except only infants with VSD or AVSD will be enrolled (no TOF). The safety profile of L-carnitine is outstanding, with no reports of toxicity from overdose reported113. In fact, the only adverse reactions reported are transient nausea and vomiting, and less commonly gastritis. However, although rare, seizures have been reported to occur in patients receiving L-carnitine. Therefore, the major adverse events that will be monitored include evidence of seizure activity and GI bleeding. As per routine, any patient suspected of having seizures is monitored with continuous EEG. Dosing is not well studied in children, particularly critically ill children67, 114-116117. In addition, the effect of CPB on L-carnitine clearance in children is not known. Therefore, a major goal of this sub-aim is to establish a pharmacokinetic profile of L-carnitine in this patient population undergoing surgery with CPB, in order to move forward with a larger randomized trial powered for efficacy in prevention of increased PVR post-bypass in at-risk infants. Plasma concentration profiles after IV bolus dosing in adults were described by a two-compartmental model67, 113, 114, 118. Usual pediatric dosing is not well delineated, but recommendations include a 50 mg/kg bolus followed by an infusion of 50mg/kg/day, that can be increased to 300 mg/kg/day113, 119. Therefore, we will begin at a lower dose (25 mg/kg), and escalate the dose after each group of 5. No intra-patient escalation will be allowed and the dose will not be escalated until all patients in the current dose level have been followed to hospital discharge or 30 days post-op and the safety and PK data have been analyzed. The DSMB will approve all dose escalations. The dosing goal will be to achieve normal or supra-normal free carnitine levels (~50 μmol/L) and low AC levels (~3 μmol/L) just before and for 24 hrs after CPB; the period with the greatest risk of pulmonary vascular morbidity.

ELIGIBILITY:
Inclusion Criteria:

* have unrestrictive VSD, AVSD
* are undergoing complete repair
* are between 2-12 months of age
* are corrected gestational age ≥34 weeks
* will have an indwelling arterial or venous line
* have not had enteral or parenteral nutrition for at least 6 hrs

Exclusion Criteria:

* have body weight < 2.0 kg
* pulmonary artery or vein abnormalities not being addressed surgically
* suspected or proven in-born error of metabolism
* have other major congenital abnormalities that affect the cardiopulmonary system
* are taking carnitine supplementation

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Blood carnitine level (free, total, and acylcarnitine) | At enrollment (first dose), and again 24 and 48 hrs after enrollment. 2 hours after enrollment (at time of second dose) and 0.5, 1.5, 3, 5, 9, 12, and 24h after the second dose.

SECONDARY OUTCOMES:
Bioavailable nitric oxide | At enrollment (first dose), and again 24 and 48 hrs after enrollment.
Plasma levels of superoxide | At enrollment (first dose), and again 24 and 48 hrs after enrollment.
Carnitine Palmityl Transporter-1 and -2 expression | At enrollment (first dose), and again 24 and 48 hrs after enrollment.
Cardiopulmonary bypass | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Echocardiographic measurements | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Estimates of PPA and right ventricular (RV) function by transesophageal ECHO (TEE)
Blood BNP level | Daily during the hospitalization, estimated to be an average of 2 weeks
Duration of mechanical ventilation | During hospitalization which is an average of 2 weeks
Vasopressor infusions | Duration of hospitalization which is an average of 2 weeks
Need for inhaled nitric oxide | During hospitalization (average of 2 weeks)
Incidence of low cardiac output syndrome | Postoperative hospitalization (average of 2 weeks)
Need for extracorporeal life support | During hospitalization (average of 2 weeks)
Plasma H202 levels | At enrollment (first dose), and again 24 and 48 hrs after enrollment.
Aortic cross clamp times | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fineman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Ghorishi Z, Milstein JM, Poulain FR, Moon-Grady A, Tacy T, Bennett SH, Fineman JR, Eldridge MW. Shear stress paradigm for perinatal fractal arterial network remodeling in lambs with pulmonary hypertension and increased pulmonary blood flow. Am J Physiol Heart Circ Physiol. 2007 Jun;292(6):H3006-18. doi: 10.1152/ajpheart.01012.2006. Epub 2007 Feb 16. PMID 17308003
- [Background] Black SM, Kumar S, Wiseman D, Ravi K, Wedgwood S, Ryzhov V, Fineman JR. Pediatric pulmonary hypertension: Roles of endothelin-1 and nitric oxide. Clin Hemorheol Microcirc. 2007;37(1-2):111-20. PMID 17641401
- [Background] Sharma S, Grobe AC, Wiseman DA, Kumar S, Englaish M, Najwer I, Benavidez E, Oishi P, Azakie A, Fineman JR, Black SM. Lung antioxidant enzymes are regulated by development and increased pulmonary blood flow. Am J Physiol Lung Cell Mol Physiol. 2007 Oct;293(4):L960-71. doi: 10.1152/ajplung.00449.2006. Epub 2007 Jul 13. PMID 17631609
- [Background] Lakshminrusimha S, Wiseman D, Black SM, Russell JA, Gugino SF, Oishi P, Steinhorn RH, Fineman JR. The role of nitric oxide synthase-derived reactive oxygen species in the altered relaxation of pulmonary arteries from lambs with increased pulmonary blood flow. Am J Physiol Heart Circ Physiol. 2007 Sep;293(3):H1491-7. doi: 10.1152/ajpheart.00185.2007. Epub 2007 May 18. PMID 17513498
- [Background] Oishi P, Sharma S, Grobe A, Azakie A, Harmon C, Johengen MJ, Hsu JH, Fratz S, Black SM, Fineman JR. Alterations in cGMP, soluble guanylate cyclase, phosphodiesterase 5, and B-type natriuretic peptide induced by chronic increased pulmonary blood flow in lambs. Pediatr Pulmonol. 2007 Nov;42(11):1057-71. doi: 10.1002/ppul.20696. PMID 17902145
- [Background] Sud N, Sharma S, Wiseman DA, Harmon C, Kumar S, Venema RC, Fineman JR, Black SM. Nitric oxide and superoxide generation from endothelial NOS: modulation by HSP90. Am J Physiol Lung Cell Mol Physiol. 2007 Dec;293(6):L1444-53. doi: 10.1152/ajplung.00175.2007. Epub 2007 Sep 7. PMID 17827253
- [Background] Oishi PE, Wiseman DA, Sharma S, Kumar S, Hou Y, Datar SA, Azakie A, Johengen MJ, Harmon C, Fratz S, Fineman JR, Black SM. Progressive dysfunction of nitric oxide synthase in a lamb model of chronically increased pulmonary blood flow: a role for oxidative stress. Am J Physiol Lung Cell Mol Physiol. 2008 Nov;295(5):L756-66. doi: 10.1152/ajplung.00146.2007. Epub 2008 Aug 29. PMID 18757524
- [Background] Sharma S, Sud N, Wiseman DA, Carter AL, Kumar S, Hou Y, Rau T, Wilham J, Harmon C, Oishi P, Fineman JR, Black SM. Altered carnitine homeostasis is associated with decreased mitochondrial function and altered nitric oxide signaling in lambs with pulmonary hypertension. Am J Physiol Lung Cell Mol Physiol. 2008 Jan;294(1):L46-56. doi: 10.1152/ajplung.00247.2007. Epub 2007 Nov 16. PMID 18024721
- [Background] Kumar S, Sun X, Sharma S, Aggarwal S, Ravi K, Fineman JR, Black SM. GTP cyclohydrolase I expression is regulated by nitric oxide: role of cyclic AMP. Am J Physiol Lung Cell Mol Physiol. 2009 Aug;297(2):L309-17. doi: 10.1152/ajplung.90538.2008. Epub 2009 May 15. PMID 19447893
- [Background] Sharma S, Kumar S, Sud N, Wiseman DA, Tian J, Rehmani I, Datar S, Oishi P, Fratz S, Venema RC, Fineman JR, Black SM. Alterations in lung arginine metabolism in lambs with pulmonary hypertension associated with increased pulmonary blood flow. Vascul Pharmacol. 2009 Nov-Dec;51(5-6):359-64. doi: 10.1016/j.vph.2009.09.005. Epub 2009 Oct 8. PMID 19818875
- [Background] Tian J, Smith A, Nechtman J, Podolsky R, Aggarwal S, Snead C, Kumar S, Elgaish M, Oishi P, Goerlach A, Fratz S, Hess J, Catravas JD, Verin AD, Fineman JR, She JX, Black SM. Effect of PPARgamma inhibition on pulmonary endothelial cell gene expression: gene profiling in pulmonary hypertension. Physiol Genomics. 2009 Dec 30;40(1):48-60. doi: 10.1152/physiolgenomics.00094.2009. Epub 2009 Oct 13. PMID 19825830
- [Background] Aggarwal S, Gross C, Fineman JR, Black SM. Oxidative stress and the development of endothelial dysfunction in congenital heart disease with increased pulmonary blood flow: lessons from the neonatal lamb. Trends Cardiovasc Med. 2010 Oct;20(7):238-46. doi: 10.1016/j.tcm.2011.11.010. PMID 22293025
- [Background] Sharma S, Kumar S, Wiseman DA, Kallarackal S, Ponnala S, Elgaish M, Tian J, Fineman JR, Black SM. Perinatal changes in superoxide generation in the ovine lung: Alterations associated with increased pulmonary blood flow. Vascul Pharmacol. 2010 Jul-Aug;53(1-2):38-52. doi: 10.1016/j.vph.2010.03.005. Epub 2010 Mar 31. PMID 20362073
- [Background] Aggarwal S, Gross CM, Kumar S, Datar S, Oishi P, Kalkan G, Schreiber C, Fratz S, Fineman JR, Black SM. Attenuated vasodilatation in lambs with endogenous and exogenous activation of cGMP signaling: role of protein kinase G nitration. J Cell Physiol. 2011 Dec;226(12):3104-13. doi: 10.1002/jcp.22692. PMID 21351102
- [Background] Sharma S, Sun X, Kumar S, Rafikov R, Aramburo A, Kalkan G, Tian J, Rehmani I, Kallarackal S, Fineman JR, Black SM. Preserving mitochondrial function prevents the proteasomal degradation of GTP cyclohydrolase I. Free Radic Biol Med. 2012 Jul 15;53(2):216-29. doi: 10.1016/j.freeradbiomed.2012.03.016. Epub 2012 Apr 16. PMID 22583703